CLINICAL TRIAL: NCT02231060
Title: Hypoxia and Outcome Prediction in Early Stage Coma: Towards an Improvement of Clinical and Electrophysiological Predictors
Brief Title: Study for the Improvement of Long-Term Outcome Prediction in Patients in Coma After Cardiac Arrest
Acronym: HOPE
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Else Kröner Fresenius Foundation (Other); University Hospital Augsburg (Other); Klinikum Ingolstadt (Other); Klinikum Rosenheim (Other); Therapiezentrum Burgau (Other); Schoen Clinic Bad Aibling (Other); Schön Klinik München Schwabing (Unknown); Asklepios Stadtklinik Bad Tölz (Unknown); Technical University of Munich (Other); Krankenhaus Barmherzige Brüder München (Unknown); Roteskreuzklinikum München (Unknown); Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Principal Investigator, Andreas Bender, Professor, Doctor Medicinae (Prof. Dr. med.), Ludwig-Maximilians - University of Munich
Other Study IDs: 2014_A55
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Anoxic-Ischemic Encephalopathy
Keywords: Outcome Prediction; Anoxic-Ischemic Encephalopathy; Coma; Vegetative State; Minimally Conscious State; Chronic Disorders of Consciousness
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Coma; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AIE after Cardiac Arrest: Male and female patients with AIE following CA.

SUMMARY:
The primary objective of HOPE is to improve the accuracy of outcome prediction in anoxic-ischemic encephalopathy following cardiac arrest by bringing under close scrutiny some of the existing methods used for this purpose (e.g. somato-sensory evoked potentials). HOPE is the first multicenter prospective cohort study on coma prognosis to control for the effect of a possible self-fulfilling prophecy at the ICU and to cover the acute and neurorehabilitation phases with a long-term follow-up longer than the usual three or six months.

DETAILED DESCRIPTION:
HOPE conducts a 2.5-year multicenter prospective cohort study in Germany on outcome prediction in the early stages of coma caused by cerebral hypoxia-ischemia.

The main features of the project are:

* Control for a self-fulfilling prophecy
* Long-term follow-up (12 months) covering acute and neurorehabilitation phases
* Use of sensitive measures of level of consciousness
* Further in-depth and systematic examination of the predictive value of somato-sensory evoked potentials (SSEP)

Using as a reference existing guidelines and previous research, we consider the following factors to be predictors of a negative outcome with a high specificity of > 90% with small 95% confidence intervals: loss of cortical N20 SEP potentials, loss of more than one brain stem reflex, non-reactive EEG, or a NSE above 33 mcg/L. We refer to the presence of any of these specific unfavourable test results during the ICU treatment as a "negative predictor". Therefore, our null hypothesis is that the probability of a favourable outcome, despite the presence of a negative predictor, is < 10%. We will use Simon's two-stage design. The null hypothesis will be tested against a one-sided alternative. In the first stage, we will accrue 72 patients. If there are 8 or fewer good outcomes in these 72 patients, the study will be discontinued because the null hypothesis could not be rejected. Otherwise, we will recruit 100 additional patients to gather a total of 172. The null hypothesis will be rejected if 28 or more favourable outcomes are observed in these 172 patients. This design yields a type I error rate of 0.05 and power of 80% if the true response rate is 25%, i.e. if indeed 25% or more patients have a favourable outcome despite a negative predictor. This calculation is based on the assumption that 25% of the enrolled patients have at least one negative predictor.

HOPE has seven data entry points (i.e. study visits).The primary endpoints are completion of the follow-up period or patient death. HOPE collects clinical and demographic data in accordance to Utstein-style recommendations. The most crucial part of the study is determining the current level of consciousness by means of the revised version of the Coma Recovery Scale (CRS-R). The CRS-R allows a precise categorization of the current level of consciousness based on a structured and systematic clinical examination of auditory, visual, motor, oromotor, communication and arousal functions. Other assessment instruments employed yield information about functional outcome/ADL, neuropsychological performance, and health-related quality of life.

Study centers will collect data prospectively following a data acquisition timeline (e.g. t0 to t6). Visits t0 to t2 will take place at acute-setting ICUs; visits t3 to t5 at neurorehabilitation centers; and visit t6 at the patients' location of residence 12 months after day 0. A manual and data dictionary will be provided to all centres along with the case report forms (CRF). All study centers will send pseudonymized data weekly by certified mail to the Central Study Centre (CSC) located at the Department of Neurology of the University of Munich. All study centres, including the CSC, will check the data for completeness, plausibility, accuracy, consistency and outliers. Legal representatives of coma patients, who decline to participate, will be asked to provide data on socio-demographic variables and reason for declining. The CSC will store the data at a database and will be responsible for safeguarding and analysing it. Patients/Legal representatives will be asked to remain in the study for a further follow-up. After completion of the follow-up period, datasets will be irreversibly anonymised.

We will analyze the positive predictive value of a dichotomous prognostic marker (favorable or unfavourable SSEP). For this purpose, we will use two definitions of favorable outcome, i.e. a functional and a behavioral one. If outcome is defined with respect to independence in daily life, we will use a modified Rankin Scale score of 0-3 (no symptoms - moderate disability, but able to walk independently) to categorize a favorable functional outcome. In the context of a catastrophic event such as cardiac arrest with high likelihood of permanent VS, it is our experience that some patients and families consider regaining functional communications skills also a favourable outcome. In a separate analysis, we will therefore use the recovery of full consciousness as measured by the CRS-R to define a favorable behavioral outcome. To analyse the effect of covariates on functional and behavioral outcomes, we will use mixed effects regression models, including both fixed and random effects. This method of analyzing longitudinal data is highly effective to examine change trajectories with several unequally spaced waves of data. Covariates will be sociodemographic variables, prognostic variables and treatment factors (e.g. use of therapeutic hypothermia), adjusted for age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Cause of admission to ICU: cardiac arrest (in or out of hospital)
* Glasgow-Coma-Scale < 9 at time of study enrolment (3 to 8 days after cardiac arrest)
* Informed consent signed by legal guardian/next-of-kin

Exclusion Criteria:

* Stroke (as it may interfere with SSEP testing)
* Pre-existing coma/vegetative state/minimally conscious state
* Terminal malignant disease
* Survival in the next 12 months extremely unlikely
* Existing advanced directive that demands cessation of therapy/life support
* Palliative care/withdrawal of life support during treatment at the ICU
* Barbiturate-induced general anesthesia during the first 3 days after cardiac arrest
* Impossibility of assessing current level of consciousness with the Glasgow Coma Scale due to a long-term deep sedation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anoxic-ischemic encephalopathy following cardiac arrest.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-10; Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Current level of consciousness as measured by the revised version of the Coma Recovery Scale (CRS-R) | There are 6 CRS-R data entry points distributed within a 12-month period, namely, 2 time points at the ICU, 3 time points during neurorehabilitation and 1 time point at the patient's residence 12 months after day 0.
  The CRS-R allows a precise categorization of the current level of consciousness based on a structured and systematic clinical examination of auditory, visual, motor, oromotor, communication and arousal functions.

SECONDARY OUTCOMES:
Regaining of functional communication skills and optimal health-related quality of life | Five data entry points distributed within a 12-month period, namely, 1 time point at the ICU, 3 time points during neurorehabilitation and 1 time point at the patient's residence 12 months after day 0.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bender, MD, Principal Investigator — Ludwig-Maximilians-Universität München
Locations (16):
- Germany (16):
  - Department of Neurology, Klinikum Augsburg, Augsburg, Bavaria
  - I. Medizinische Klinik, Klinikum Augsburg, Augsburg, Bavaria
  - Schön Klinik Bad Aibling, Bad Aibling, Bavaria
  - Dept of Neurology, Asklepios Stadtklinik Bad Tölz, Bad Tölz, Bavaria
  - Therapiezentrum Burgau, Burgau, Bavaria
  - Medizinische Klinik I und IV, Klinikum Ingolstadt, Ingolstadt, Bavaria
  - Neurologische Klinik, Klinikum Ingolstadt, Ingolstadt, Bavaria
  - Deutsches Herzzentrum Muenchen, Munich, Bavaria
  - Krankenhaus Barmherzige Brüder München, Munich, Bavaria
  - Schön Klinik München Schwabing, Munich, Bavaria
  - Department of Neurology, University of Munich, Munich, Bavaria
  - Internal ICU, Medical Clinic and Polyclinic IV, University of Munich, Munich, Bavaria
  - Medizinische Klinik und Poliklinik I, University of Munich, Munich, Bavaria
  - Department of Neurology, Munich, Bavaria
  - Clinic for Anesthesiology, University of Munich, Munich, Bavaria
  - Neurologische Klinik, RoMed Klinikum Rosenheim, Rosenheim, Bavaria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lopez-Rolon A, Bender A; Project HOPE Investigator Group. Hypoxia and Outcome Prediction in Early-Stage Coma (Project HOPE): an observational prospective cohort study. BMC Neurol. 2015 May 15;15:82. doi: 10.1186/s12883-015-0337-x. PMID 25971341
- See also: Hypoxia and Outcome Prediction in Early-Stage Coma (Project HOPE): an observational prospective cohort study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4451883/